CLINICAL TRIAL: NCT00894153
Title: Open-Label, Multi-Center, Randomized, Active-Controlled, Phase 4 Study of rAd-p53 Gene Therapy Combined With Chemotherapy and Radiotherapy in Treament of Head and Neck Cancer in Advanced Stage
Brief Title: p53 Gene Therapy for Head and Neck Malignant Tumors in Advanced Stage
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen SiBiono GeneTech Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: rAd-p53-001
Record Dates: First submitted 2009-05-04; First posted 2009-05-06 (Estimated); Last update posted 2012-04-09 (Estimated); Status verified 2010-02

CONDITIONS: Neoplasms
Keywords: p53 gene; head and neck malignent tumors; gene therapy
MeSH Terms: conditions — Neoplasms | interventions — Drug Therapy; Genes, p53; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- chemo plus p53 (Experimental): chemotherapy plus p53
  Interventions: Drug: chemotherapy plus p53
- chemo only (Active Comparator): chemotherapy group
  Interventions: Drug: chemotherapy
- radio (Active Comparator): radiotherapy
  Interventions: Radiation: radiotherapy

INTERVENTIONS:
Drug: chemotherapy plus p53 — chemotherapy plus p53
  Arms: chemo plus p53
Drug: chemotherapy — chemotherapy
  Arms: chemo only
Radiation: radiotherapy — radiotherapy
  Arms: radio

SUMMARY:
This is multicenter, open-label, randomized, active-controled, phase IV study of local direct intra-tumor injection of rAd-p53 monotherapy, with concurrent chemotherapy , with concurrent radiotherapy, or combination with surgery for treatment of head and neck malignant tumors in advanced stage .

DETAILED DESCRIPTION:
Primary objectives of this study is to determine the efficacy profiles of rAd-p53 intra-tumor injection alone, with concurrent chemotherapy, with concurrent radiotherapy, or combination with surgery for treatment of head and neck malignant tumors in advanced stage (stage III or IV) including target lesion complete response rate (LCR) and overall target lesion response rate (OLR), response duration (RD), and progress-free survival (PFS).

The secondary objectives of this study is to investigate overall response rate (OPCR) and overall complete response rate (OCR), overall survival (OS), ECOG, and safety of rAd-p53 monotherapy and combined with chemotherapy, radiotherapy or surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Advanced stages of head and neck malignant tumors (stage III and VI)
2. At least one target tumor can be injected with study drug, the largest diameter greater than 2 cm
3. Histologically confirmed head and neck malignant tumors
4. No prior chemotherapy, radiotherapy or biological tumor therapy in 2 weeks
5. Age: 18-85 years old
6. Expected to survive more 12 weeks
7. ECOG:0-2
8. Neutrophils≥1.5×109/L,Platelet≥ 80×109/L, Hb≥80g/L, bilitubin≤2mg/dl,ALT and AST ≤2×institutional upper limit of normal, Cr ≤1.5×institutional upper limit of normal,coagulation tests (PTT and INR) within normal range
9. Subject provided signed informed consent

Exclusion Criteria:

1. Hypersensitive to study drug
2. Tumor(s) locate very close to important blood vessels and nerves, which affect injection
3. With a coagulation and bleeding disorder
4. With uncontrolled, intercurrent illness including but limited to symptomatic neurological illness, symptomatic congestive heart failure, unstable angina pectoris, significant pulmonary disease or hypoxia, or psychiatric illness
5. Local infection close to injection site or systemic infection
6. Pregnant or lactating
7. Principle investigator consider not suitable

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2009-05; Primary Completion 2012-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Efficacy | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of oral and maxillofacial surgery, Huaxi university of medical science, Chendu, Shichuan, China